CLINICAL TRIAL: NCT02558283
Title: A Safety and Efficacy Study of JUVÉDERM® VOLIFT® With Lidocaine and Restylane® for Nasolabial Folds in Chinese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: VOLIFT-002
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Nasolabial Fold

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JUVÉDERM® VOLIFT® with Lidocaine - Right Side (Experimental): JUVÉDERM® VOLIFT® with lidocaine injected into the right nasolabial fold on Day 1, with optional touch-up injections into the right nasolabial fold on Month 1.
  Interventions: Device: JUVÉDERM® VOLIFT® with Lidocaine
- Restylane® - Right Side (Active Comparator): Restylane® injected into the right nasolabial fold on Day 1, with optional touch-up injections into the right nasolabial fold on Month 1.
  Interventions: Device: Restylane®
- JUVÉDERM® VOLIFT® with Lidocaine - Left Side (Experimental): JUVÉDERM® VOLIFT® with lidocaine injected into the left nasolabial fold on Day 1, with optional touch-up injections into the left nasolabial fold on Month 1.
  Interventions: Device: JUVÉDERM® VOLIFT® with Lidocaine
- Restylane® - Left Side (Active Comparator): Restylane® injected into the left nasolabial fold on Day 1, with optional touch-up injections into the left nasolabial fold on Month 1.
  Interventions: Device: Restylane®

INTERVENTIONS:
Device: JUVÉDERM® VOLIFT® with Lidocaine — JUVÉDERM® VOLIFT® with lidocaine injected into the nasolabial fold on Day 1, with optional touch-up injections into the nasolabial fold on Month 1.
  Arms: JUVÉDERM® VOLIFT® with Lidocaine - Left Side; JUVÉDERM® VOLIFT® with Lidocaine - Right Side
Device: Restylane® — Restylane® injected into the nasolabial fold on Day 1, with optional touch-up injections into the nasolabial fold on Month 1.
  Arms: Restylane® - Left Side; Restylane® - Right Side

SUMMARY:
This is a safety and efficacy study of JUVÉDERM® VOLIFT® with Lidocaine and Restylane® in Chinese adults with nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

* Presence of nasolabial folds
* Agree to refrain from treatment with other anti-wrinkle/volumizers below the eye for the duration of the study

Exclusion Criteria:

* Ever received semi-permanent fillers or permanent facial implants below the eyes, or plans to receive these treatments during the study
* Undergone temporary dermal filler treatment (eg, hyaluronic acid or collagen) below the eyes within 12 months, or plans to undergo these treatments during the study
* Undergone facial tissue augmentation with fat injections, botulinum toxin injections, mesotherapy, or cosmetic facial procedures in the face or neck within 6 months, or plans to undergo these treatments during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Investigator's Assessment of Severity of Each Nasolabial Fold (NLF) on the 5-Point NLF Severity Scale (NLFSS) | Month 6

SECONDARY OUTCOMES:
Subject's Assessment of Procedural Pain on an 11-Point Scale | Day 1
Investigator's Assessment of Each NLF on the 5-Point Global Aesthetic Improvement Scale (GAIS) | Month 6
Subject's Assessment of Each NLF on the 5-Point GAIS | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Yi Jia, Study Director — Allergan
Locations (5):
- China (5):
  - China Japan Friendship Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - General Hospital of Guangzhou Military Command of PLA, Guangzhou
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Guangzhou
  - Shanghai 9th Hospital, Shanghai